CLINICAL TRIAL: NCT05434182
Title: Groin Surgical Site Infection Incidence in Vascular Surgery With Intradermal Suture Versus Metallic Stapling Skin Closure: A Pragmatic Open-Label Parallel-Group Randomized Clinical Trial
Brief Title: Intradermal Suture Versus Stapling for Groin Skin Closure in Vascular Surgery (VASC-INF Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Albert Gonzalez-Sagredo, Surgeon at the Vascular Surgery and Angiology Department, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VASC-INF-2021-01
Record Dates: First submitted 2022-06-16; First posted 2022-06-27 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Surgical Site Infection
Keywords: Femoral approach; Intradermal suture; Metallic staples; Surgical Site Infection; Groin
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intradermal Suture Group (Experimental): Vascular surgery patients undergoing a femoral approach surgery and randomized to this group will have their skin closed with an intradermal suture using Monosyn® (Braun®) 4/0 absorbable monofilament.
  Interventions: Procedure: Intradermal Suture
- Metallic Staples (Active Comparator): Vascular surgery patients undergoing a femoral approach surgery and randomized to this group will have their skin closed with metallic stapling using Visistat® (Weck®) 35W skin stapler.
  Interventions: Procedure: Metallic Staples

INTERVENTIONS:
Procedure: Intradermal Suture — Skin closure with an intradermal suture using Monosyn® (Braun®) 4/0 absorbable monofilament.
  Arms: Intradermal Suture Group
Procedure: Metallic Staples — Skin closure with metallic stapling using Visistat® (Weck®) 35W skin stapler.
  Arms: Metallic Staples

SUMMARY:
Surgical site infection (SSI) is one of the most frequent and fearsome complications in vascular surgery due to its high morbidity and mortality. In addition, SSI is one of the factors related to the development of prosthetic infection. Consequently, it represents a significant increase in hospital stay and healthcare costs.

A 2021 meta-analysis on groin SSI prevention strategies in arterial surgeries reported that using intradermal sutures could be associated with a lower SSI rate. The published results from a single-center retrospective study comparing SSI rates before and after implementing an SSI prevention protocol also suggest better outcomes with intradermal suturing.

This study aims to assess the SSI incidences of both skin closure techniques in vascular surgery patients undergoing femoral artery approach through a perpendicular groin skin incision.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic lower limb ischemia or aortic, iliac, or femoral aneurysm
* With a scheduled surgery for one of the following indications:
* Femoropopliteal Bypass
* Femorodistal Bypass
* Aortobifemoral Bypass
* Axillofemoral or Axillobifemoral Bypass
* Femorofemoral Bypass
* Femoral Endarterectomy
* Femoral approach for exclusion of an aortic aneurysm
* Surgical procedure with an incision perpendicular to the inguinal fold
* Patients who undergo both unilateral and bilateral surgical approaches *

  *Note: We will consider one patient as one intervention (i.e., bilateral approaches will be quantified as one single inguinal surgical approach). In the case of bilateral procedures, the same closure technique will be used for both sides.
* Patients who sign the written informed consent

Exclusion Criteria:

* Background of a previous surgical intervention in the groin area.
* Femoral approach carried out in a surgical emergency setting
* Femoral approach performed due to a femoral pseudoaneurysm
* A surgical procedure performed with a transverse/oblique incision to the groin
* A patient who withdraws consent for participating in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Number (percentage) of patients who present a femoral approach SSI* -(superficial and/or deep) up to 28 (±2) after surgery. | 28 (±2) days after surgery
  According to the National Healthcare Safety Network (NHSN) Classification

SECONDARY OUTCOMES:
Number (percentage) of patients with other surgical wound complications up to 28 (±2) days after surgery. | 28 (±2) days after surgery
  Complications include but are not limited to seroma, hematoma, lymphorrhagia.
Number (percentage) of patients who develop sepsis up to 28 (±2) days after surgery | 28 (±2) days after surgery
Number (percentage) of patients with SSI who develop sepsis up to 28 (±2) days after surgery. | 28 (±2) days after surgery
Time of prophylactic antibiotic administration | 28 (±2) days after surgery
Types of microorganisms isolated from skin microbiological culture, subcutaneous tissue sample culture, and SSI secretion culture up to 28 (±2) days after surgery. | 28 (±2) days after surgery
Types of antibiotic therapy used in patients with SSI | 84 (±7) days after surgery
Plasma albumin concentration | Baseline visit to 28 (±2) days after surgery
Body Mass Index | Baseline visit to 28 (±2) days after surgery
Surgical incision length | On the day of performing the surgical procedure
  Length (in centimeters [cm]) of the cutaneous incision performed to gain access to the surgical site. This information will be collected on the day of performing the surgery, once it is over.
Total surgery duration | On the day of performing the surgical procedure
  Duration (in minutes) of the surgical procedure. This information will be collected on the day of performing the surgery, once it is over.
Type of hemostatic material used during surgery | On the day of performing the surgical procedure
  This information will be collected on the day of performing the surgery, once it is over.
Number of days between hospital admission and the surgical intervention | From the day of hospital admission to the day of performing the surgical procedure
  The number of days gone by from hospital admission until the day the surgery is performed. This information will be collected on the day of performing the surgery, once it is over.
Number (percentage) of patients who present a femoral approach SSI (superficial and/or deep) up to 84 (±7) days after surgery | 84 (±7) days after surgery
  According to the NHSN classification

CONTACTS AND LOCATIONS:
Overall Officials: Elena Iborra, M.D., Ph.D., Principal Investigator — Hospital Universitari de Bellvitge - Angiology and Vascular Surgery Department
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The sponsor will oversee the dataset. Granting access to this information will be evaluated on a case-by-case basis and upon reasonable request by the interested party.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Perencevich EN, Sands KE, Cosgrove SE, Guadagnoli E, Meara E, Platt R. Health and economic impact of surgical site infections diagnosed after hospital discharge. Emerg Infect Dis. 2003 Feb;9(2):196-203. doi: 10.3201/eid0902.020232. PMID 12603990
- [Background] Chakfe N, Diener H, Lejay A, Assadian O, Berard X, Caillon J, Fourneau I, Glaudemans AWJM, Koncar I, Lindholt J, Melissano G, Saleem BR, Senneville E, Slart RHJA, Szeberin Z, Venermo M, Vermassen F, Wyss TR, Esvs Guidelines Committee, de Borst GJ, Bastos Goncalves F, Kakkos SK, Kolh P, Tulamo R, Vega de Ceniga M, Document Reviewers, von Allmen RS, van den Berg JC, Debus ES, Koelemay MJW, Linares-Palomino JP, Moneta GL, Ricco JB, Wanhainen A. Editor's Choice - European Society for Vascular Surgery (ESVS) 2020 Clinical Practice Guidelines on the Management of Vascular Graft and Endograft Infections. Eur J Vasc Endovasc Surg. 2020 Mar;59(3):339-384. doi: 10.1016/j.ejvs.2019.10.016. Epub 2020 Feb 5. No abstract available. PMID 32035742
- [Background] Groin wound Infection after Vascular Exposure (GIVE) Study Group. Groin wound infection after vascular exposure (GIVE) multicentre cohort study. Int Wound J. 2021 Apr;18(2):164-175. doi: 10.1111/iwj.13508. Epub 2020 Nov 25. PMID 33236858
- [Background] Kirkland KB, Briggs JP, Trivette SL, Wilkinson WE, Sexton DJ. The impact of surgical-site infections in the 1990s: attributable mortality, excess length of hospitalization, and extra costs. Infect Control Hosp Epidemiol. 1999 Nov;20(11):725-30. doi: 10.1086/501572. PMID 10580621
- [Background] Gwilym BL, Dovell G, Dattani N, Ambler GK, Shalhoub J, Forsythe RO, Benson RA, Nandhra S, Preece R, Onida S, Hitchman L, Coughlin P, Saratzis A, Bosanquet DC. Editor's Choice - Systematic Review and Meta-Analysis of Wound Adjuncts for the Prevention of Groin Wound Surgical Site Infection in Arterial Surgery. Eur J Vasc Endovasc Surg. 2021 Apr;61(4):636-646. doi: 10.1016/j.ejvs.2020.11.053. Epub 2021 Jan 7. PMID 33423912
- [Background] Nikulainen V, Helmio P, Hurme S, Hakovirta H. Intra-Dermal Absorbable Suture in the Groin Incision Associated with Less Groin Surgical Site Infections than Trans-Dermal Sutures in Vascular Surgical Patients. Surg Infect (Larchmt). 2019 Jan;20(1):45-48. doi: 10.1089/sur.2018.202. Epub 2018 Oct 6. PMID 30300081
- [Background] Parizh D, Ascher E, Raza Rizvi SA, Hingorani A, Amaturo M, Johnson E. Quality improvement initiative: Preventative Surgical Site Infection Protocol in Vascular Surgery. Vascular. 2018 Feb;26(1):47-53. doi: 10.1177/1708538117719155. Epub 2017 Jul 14. PMID 28708024
- [Background] Engin C, Posacioglu H, Ayik F, Apaydin AZ. Management of vascular infection in the groin. Tex Heart Inst J. 2005;32(4):529-34. PMID 16429897
- [Background] Yashar JJ, Weyman AK, Burnard RJ, Yashar J. Survival and limb salvage in patients with infected arterial prostheses. Am J Surg. 1978 Apr;135(4):499-504. doi: 10.1016/0002-9610(78)90027-2. PMID 637195
- [Background] Pleger SP, Nink N, Elzien M, Kunold A, Koshty A, Boning A. Reduction of groin wound complications in vascular surgery patients using closed incision negative pressure therapy (ciNPT): a prospective, randomised, single-institution study. Int Wound J. 2018 Feb;15(1):75-83. doi: 10.1111/iwj.12836. Epub 2017 Oct 25. PMID 29068153
- [Background] Antonios VS, Noel AA, Steckelberg JM, Wilson WR, Mandrekar JN, Harmsen WS, Baddour LM. Prosthetic vascular graft infection: a risk factor analysis using a case-control study. J Infect. 2006 Jul;53(1):49-55. doi: 10.1016/j.jinf.2005.10.004. Epub 2005 Nov 28. PMID 16310254
- [Background] Oderich GS, Panneton JM. Aortic graft infection. What have we learned during the last decades? Acta Chir Belg. 2002 Feb;102(1):7-13. doi: 10.1080/00015458.2002.11679254. No abstract available. PMID 11925745
- [Background] Siracuse JJ, Nandivada P, Giles KA, Hamdan AD, Wyers MC, Chaikof EL, Pomposelli FB, Schermerhorn ML. Prosthetic graft infections involving the femoral artery. J Vasc Surg. 2013 Mar;57(3):700-5. doi: 10.1016/j.jvs.2012.09.049. Epub 2013 Jan 9. PMID 23312940
- [Background] Wiseman JT, Fernandes-Taylor S, Barnes ML, Saunders RS, Saha S, Havlena J, Rathouz PJ, Kent KC. Predictors of surgical site infection after hospital discharge in patients undergoing major vascular surgery. J Vasc Surg. 2015 Oct;62(4):1023-1031.e5. doi: 10.1016/j.jvs.2015.04.453. Epub 2015 Jul 3. PMID 26143662
- [Background] Leekha S, Lahr BD, Thompson RL, Sampathkumar P, Duncan AA, Orenstein R. Preoperative risk prediction of surgical site infection requiring hospitalization or reoperation in patients undergoing vascular surgery. J Vasc Surg. 2016 Jul;64(1):177-84. doi: 10.1016/j.jvs.2016.01.029. Epub 2016 Feb 27. PMID 26926939
- [Background] Pounds LL, Montes-Walters M, Mayhall CG, Falk PS, Sanderson E, Hunter GC, Killewich LA. A changing pattern of infection after major vascular reconstructions. Vasc Endovascular Surg. 2005 Nov-Dec;39(6):511-7. PMID 16382265
- [Background] Gurusamy KS, Toon CD, Allen VB, Davidson BR. Continuous versus interrupted skin sutures for non-obstetric surgery. Cochrane Database Syst Rev. 2014 Feb 14;2014(2):CD010365. doi: 10.1002/14651858.CD010365.pub2. PMID 24526375
- [Derived] Gonzalez-Sagredo A, Gil Olaria M, D'Oria M, Lopez-Garcia P, Grando B, Gonzalo Villanueva B, Espinar Garcia E, Carnaval T, Llagostera S, Lepidi S, Vila R, Iborra E, Videla S. Randomized clinical trial of intradermal suture and metallic stapling for incisional groin closure after vascular surgery (VASC-INF trial). Br J Surg. 2025 Nov 6;112(11):znaf256. doi: 10.1093/bjs/znaf256. PMID 41289050
- [Derived] Correia RM, Nakano LC, Vasconcelos V, Cristino MA, Flumignan RL. Prevention of infection in peripheral arterial reconstruction of the lower limb. Cochrane Database Syst Rev. 2025 Oct 29;10(10):CD015022. doi: 10.1002/14651858.CD015022.pub2. PMID 41159585
- [Derived] Cristino MA, Nakano LC, Vasconcelos V, Correia RM, Flumignan RL. Prevention of infection in aortic or aortoiliac peripheral arterial reconstruction. Cochrane Database Syst Rev. 2025 Apr 22;4(4):CD015192. doi: 10.1002/14651858.CD015192.pub2. PMID 40260835

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT05434182/Prot_SAP_000.pdf